CLINICAL TRIAL: NCT07172204
Title: The Efficacy and Safety of VA Alternating With Low-dose CHA in the Treatment of Newly Diagnosed Unfit AML: a Prospective, Multi-centers, Single Arm Phase II Study
Brief Title: Alternating Regimen of VA and Low-dose CHA in the Treatment of Unfit Newly Diagnosed AML
Acronym: CHANCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Jie Sun, Principle Attending, Associated Professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250072C
Record Dates: First submitted 2025-08-19; First posted 2025-09-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Intensive Chemotherapy Unfit; Newly Diagnosed Acute Myeloid Leukemia (AML); Age ≥60
Keywords: Acute Myeloid Leukemia; Venetoclax; alternating; Homoharringtonine; Cladribine; age 60 and older; intensive chemotherapy unfit; newly diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VA alternating with low-CHA (Experimental): single treatment arm
  Interventions: Drug: Alternately treated with VA/low CHA regimen

INTERVENTIONS:
Drug: Alternately treated with VA/low CHA regimen — 1. Induction Phase (4 alternating cycles):
     Participants will receive 4 cycles of alternating therapy:
     * VA Cycle:
       * Venetoclax 400 mg PO daily on Days 1-28
       * Azacitidine 75 mg/m² SC daily on Days 1-7
     * Low-dose CHA Cycle:
       * Cladribine 5 mg/m² IV daily on Days 1-3
       * Homoharringtonine 1 mg/m² IV daily on Days 1-5
       * Cytarabine 20 mg SC every 12 hours on Days 1-10 Alternating sequence: VA → CHA → VA → CHA → VA → CHA → VA → CHA
  2. Maintenance Phase (24 months):
  Following induction, participants will receive:
  * Venetoclax 400 mg PO daily on Days 1-28
  * Azacitidine 75 mg/m² SC daily on Days 1-7 Repeated every 28 days for 24 cycles.
  We aimed to compare this clinical intervention with standard VA which is:
  * Venetoclax 400 mg PO daily on Days 1-28
  * Azacitidine 75 mg/m² SC daily on Days 1-7 Repeated every 28 days for at least 24 cycles.

SUMMARY:
This phase II trial tests how well VA alternating with low-dose CHA works in treating unfit patients with newly diagnosed acute myeloid leukemia (AML). This is a prospective, multi-centers, single arm phase II study aimed to overcome VEN resistance and achieve greater MRD negative rate, providing better control of treatment for unfit AML.

DETAILED DESCRIPTION:
This clinical study protocol investigates a novel treatment for newly diagnosed Acute Myeloid Leukemia (AML) patients ineligible to receive intensive chemotherapy (IC). Eligibility is defined as age ≥60 or age 18-59 with significant comorbidities. Key exclusions include specific AML subtypes including Acute promyelocytic leukemia (APL); FLT3-ITD mutations and active infections. The Intervention is a two-phase regimen. The Induction Phase consists of four alternating 28-day cycles of Venetoclax + Azacitidine (VA) and low-dose Cladribine + Homoharringtonine + Cytarabine (CHA). This is followed by a Maintenance Phase of 24 cycles of VA therapy. The Primary Endpoint is the rate of Minimal Residual Disease (MRD) negativity after two alternating cycles. Secondary Endpoints include composite complete remission rate, overall survival, and incidence of treatment-emergent adverse events. Clear Withdrawal Criteria are defined for situations involving unacceptable toxicity, lack of therapeutic benefit, or patient/investigator decision.

ELIGIBILITY:
Inclusion Criteria:

* Understand the research and sign a written informed consent form;
* Be newly diagnosed with AML according to WHO 2022 criteria without prior treatment;
* or unwilling to undergo IC. Ineligibility for IC is defined as meeting any of the following criteria:
* Age ≥ 60 years
* Age 18-59 years but ineligible for intensive chemotherapy (IC) , meet ≥1 of the following:

  * Eastern Cooperative Oncology Group (ECOG) performance status ≥2 at screening;
  * Severe heart failure (congestive heart failure requiring treatment or myocardial infarction history with ejection fraction ≤50%);
  * Severe pulmonary dysfunction (DLCO ≤65%, FEV1 ≤65%, dyspnea at rest, or oxygen dependence);
  * Severe renal insufficiency requiring dialysis;
  * Child-Pugh B or C cirrhosis, or hepatic impairment with total bilirubin >1.5×ULN;
* Mental illness requiring inpatient psychiatric treatment;
* Any comorbidity deemed by physician to contraindicate IC.

Exclusion Criteria:

* Diagnosis of: AML arising from chronic myeloid leukemia (CML); myeloid sarcoma; acute promyelocytic leukemia (APL) or presence of FLT3-ITD mutations;
* Active malignancies (except adequately treated carcinoma in situ or basal cell carcinoma) within 2 years prior to Cycle 1 Day 1 (C1D1);
* Major surgery or systemic anticancer therapy within 28 days before C1D1;
* Known hypersensitivity to: Active pharmaceutical ingredients: cladribine, homoharringtonine, cytarabine, venetoclax, azacitidine; Any excipients in study drug formulations;
* GI conditions impairing oral drug absorption: Dysphagia; short-gut syndrome; gastroparesis or related disorders;
* Uncontrolled active infection;
* Controlled infection permitted if: Afebrile (<38°C) and hemodynamically stable (SBP >90 mmHg, HR <100 bpm) for ≥72 hours pre-C1D1; on non-interacting antimicrobial regimen; active HBV/HCV infection (Chronic carriers require PI approval with viral load monitoring); HIV-positive patients receiving HAART;
* Pregnancy/lactation or refusal of contraception: Negative serum β-hCG within 24h pre-C1D1;
* Psychiatric disorders or social circumstances compromising protocol compliance;
* Prior AML-directed therapy except: cytoreduction for hyperleukocytosis per institutional guidelines (hydroxyurea, leukapheresis); supportive growth factors;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Negative rate of minimal residual lesions (MRD) | At day28 of the second alternating (one alternating is VA plus low-CHA)
  Proportion of patients achieving MRD-negative status (≤0.1% leukemic blasts by flow cytometry) after two cycles of alternating VA/CHA therapy

SECONDARY OUTCOMES:
composite complete remission, CRc | At day28 of the first alternating and the second alternating (one alternating is VA plus low-CHA)
  Proportion achieving CR or CRi per ELN 2022 criteria at each cycle completion
Overall response rate, ORR | At day28 of the first alternating and the second alternating (one alternating is VA plus low-CHA)
  Proportion achieving PR or better (CR/CRh/CRi/MLFS/PR) per IWG criteria at each cycle completion
Overall Survival, OS | Time from enrollment to death from any cause, whichever came first, assessed up to 24 months
  Time from enrollment to death from any cause, whichever came first (censored at last follow-up for survivors)
disease-free survival, DFS | From the date of first response until the date of relapse or death from any cause, whichever came first, assessed up to 24 months
  Time from first response to relapse or death (censored at last disease assessment)
MRD negative DFS, DFS-MRD | From the date of first MRD-negative status until the date of MRD-positive, relapse or death due to relapse, whichever came first, assessed up to 24months.
  Time from first MRD-negative status to MRD-positive (confirmed by a second check within 2 weeks).
Event-free survival, EFS | from enrollment until the date of treatment failure, relapse or death from any cause, whichever came first, assessed up to 24 months
  Time from enrollment to treatment failure (not achieved PR after the first alternating, or not achieved CR after 2 alternatings, or continuous MRD positive after 4 alternatings), relapse, or death. （one alternating is VA plus low-CHA)
Incidence of adverse events (AEs) | up to 3 years
  Incidence of CTCAE v6.0-graded AEs from day 1 of treatment to study completion

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dr. Sun, M.D, Ph.D, Principal Investigator — Bone Marrow Transplantation Center of The First Affiliated Hospital, Zhejiang University School of Medicine; Shanshan Prof. Pei, Ph.D, Study Director — Liangzhu Laboratory, Zhejiang University School of Medicine
Locations (5):
- China (5):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shenzhen University General Hospital, Shenzhen, Guangdong
  - the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - the Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Bone Marrow Transplantation Center, the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared from the date of publication to 6 months after.
Access Criteria: Contact the team by e-mail or other specified contact information described on publication